CLINICAL TRIAL: NCT01202227
Title: An Open-Label Long-Term Study Of Pregabalin For The Treatment Of Central Neuropathic Pain (Post Spinal Cord Injury Pain, Post Stroke Pain, And Multiple Sclerosis Pain)
Brief Title: An Open-Label Long-Term Study Of Pregabalin For The Treatment Of Central Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081252
Record Dates: First submitted 2010-08-31; First posted 2010-09-15 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2013-04

CONDITIONS: Spinal Cord Diseases; Spinal Cord Injuries; Neuralgia; Pain
Keywords: Central Nervous System Diseases; Therapeutic Uses; Wounds and Injuries; Trauma; Nervous System; pregabalin
MeSH Terms: conditions — Spinal Cord Diseases; Spinal Cord Injuries; Neuralgia; Pain; Central Nervous System Diseases; Wounds and Injuries; Neurologic Manifestations | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregabalin (Experimental): Flexible dosing in 4 weeks followed by 48 weeks maintenance and one week taper period
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: pregabalin — Pregabalin capsules taken twice a daily (150-600mg/day)

SUMMARY:
The purpose of this study is to assess the safety of the long-term use of pregabalin at doses up to 600 mg/day in patients with central neuropathic pain (post spinal cord injury pain, post stroke pain, and multiple sclerosis pain).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for subjects to be shifted from Study A0081107

* Subjects who completed the 18-week study period in Study A0081107 conducted for chronic neuropathic pain after spinal cord injury;
* Subjects who completed assessments of all efficacy endpoints until the end of the treatment phase of the preceding Study A0081107 (V7);

Inclusion criteria for subjects to be new participants in this study

* Subjects with central neuropathic pain after stroke or multiple sclerosis;
* At least 6 months have passed after the onset of central neuropathic pain;
* Pain VAS at least 40mm in Visit 1 and Visit 2;

Exclusion Criteria:

* Creatinine clearance < 60 mL/min;
* Platelet count < 100 × 103/mm3 ; White blood cell (WBC) count < 2500 / mm3; Neutrophil count < 1500/ mm3;
* Subjects who are expected to require surgery during the trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- Japan (26):
  - Chubu Rosai Hospital, Nagoya, Aichi-ken
  - Kimura Clinic, Nagoya, Aichi-ken
  - Nagoya Kyoritsu Clinic, Nagoya, Aichi-ken
  - Senboku Kumiai General Hospital, Daisen, Akita
  - Go neurosurgical clinic, Chikushi-gun, Fukuoka
  - Spinal Injuries Center, Iizuka, Fukuoka
  - Brain Attack Center Ota Memorial Hospital, Fukuyama, Hiroshima
  - Hokkaido Chuo Rosai Hospital Sekison Center, Bibai, Hokkaido
  - Hakodate Central General Hospital, Hakodate, Hokkaido
  - Kobe Tokushukai Hospital, Kobe, Hyōgo
  - Aida Kinen Rehabilitation Hospital, Moriya, Ibaraki
  - General Hanamaki Hospital, Hanamaki, Iwate
  - Uchida Rehabilitation Orthopedic Clinic, Kawasaki, Kanagawa
  - Kumamoto Rehabilitation Hospital, Kikuchi-gun, Kumamoto
  - Kohnan Hospital, Sendai, Miyagi
  - Sendai Pain Clinic, Sendai, Miyagi
  - National Hospital Organization Niigata National Hospital, Kashiwazaki, Niigata
  - Nakamura Hospital, Beppu, Oita Prefecture
  - Kitasato University Kitasato Institute Medical Center Hospital, Kitamoto, Saitama
  - Kamitsuga General Hospital, Kanuma, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Jukoukai hospital, Koto-ku, Tokyo
  - National Hospital Organization, Murayama Medical Center, Musashimurayama-shi, Tokyo
  - Okitama Public General Hospital, Higashiokitama-gun, Yamagata
  - Tokushima University Hospital, Tokushima
  - National Hospital Organization Yamagata Hospital, Yamagata

REFERENCES:
- [Derived] Onouchi K, Koga H, Yokoyama K, Yoshiyama T. An open-label, long-term study examining the safety and tolerability of pregabalin in Japanese patients with central neuropathic pain. J Pain Res. 2014 Jul 28;7:439-47. doi: 10.2147/JPR.S63028. eCollection 2014. PMID 25114584
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081252&StudyName=An%20Open-Label%20Long-Term%20Study%20Of%20Pregabalin%20For%20The%20Treatment%20Of%20Central%20Neuropathic%20Pain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese patients with central neuropathic pain after spinal cord injury who had completed the preceding A0081107 study (NCT00407745) were eligible for this study, and Japanese patients with pain after cerebral stroke or with multiple sclerosis pain were newly recruited.
Pre-assignment Details: Participants who had joined A0081107 study (NCT00407745) were treated with pregabalin or placebo for 16 weeks and underwent tapering phase prior to this study.
Groups:
- Pregabalin: Study period consisted of 4-week dose adjustment phase followed by 48-week maintenance and one-week tapering phase. All participants were given pregabalin twice a day (BID) in the morning and evening. Participants first received 75 milligram (mg) of pregabalin in the evening of Day 1, and then 150 mg/day from Day 2 onward during the first week. The dosage could be adjusted to the maintenance dose of 150, 300, 450, or 600 mg/day by one step (±150 mg/day) in consideration of safety and efficacy on pain control during the dose adjustment phase.
Period: Overall Study
Arm/Group | Pregabalin
Started | 103 (Treated)
Completed | 84
Not Completed | 19
Not completed — Adverse Event | 16
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Age, Customized [Number; unit: Participants]
  >=18 and <45 years | 15
  >= 45 and <65 years | 60
  >=65 years | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Peripheral Edema
Description: Number of participants who had peripheral edema in lower extremities. Edema was categorized as follows: trace, pitting 1 (lower leg), 2 (lower leg to knee), and 3 (above knee and /or presacral edema).
Time Frame: Baseline, Weeks 4, 20, 36, 52, and 53
Population: The safety analysis set consists of all participants who received at least one dose of study medication in this long-term study.
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Participants
  Trace at Baseline (n=103) | 5
  Pitting +1 at Baseline (n=103) | 9
  Pitting +2 at Baseline (n=103) | 2
  Pitting +3 at Baseline (n=103) | 0
  Trace at Week 4 (n=101) | 8
  Pitting +1 at Week 4 (n=101) | 8
  Pitting +2 at Week 4 (n=101) | 4
  Pitting +3 at Week 4 (n=101) | 1
  Trace at Week 20 (n=93) | 8
  Pitting +1 at Week 20 (n=93) | 3
  Pitting +2 at Week 20 (n=93) | 7
  Pitting +3 at Week 20 (n=93) | 0
  Trace at Week 36 (n=90) | 14
  Pitting +1 at Week 36 (n=90) | 7
  Pitting +2 at Week 36 (n=90) | 3
  Pitting +3 at Week 36 (n=90) | 0
  Trace at Week 52/early termination (n=100) | 10
  Pitting +1 at Week 52/early termination (n=100) | 7
  Pitting +2 at Week 52/early termination (n=100) | 2
  Pitting +3 at Week 52/early termination (n=100) | 0
  Trace at Week 53/early termination (n=78) | 9
  Pitting +1 at Week 53/early termination (n=78) | 5
  Pitting +2 at Week 53/early termination (n=78) | 0
  Pitting +3 at Week 53/early termination (n=78) | 0

2. Primary Outcome: Number of Participants With Facial/Periorbital Edema
Description: Number of participants who had facial or periorbital edema.
Time Frame: Baseline, Weeks 4, 20, 36, 52, and 53
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Participants
  Baseline (n=103) | 0
  Week 4 (n=101) | 0
  Week 20 (n=93) | 0
  Week 36 (n=90) | 0
  Week 52/early termination (n=100) | 1
  Week 53/early termination (n=78) | 0

3. Primary Outcome: Number of Participants With Generalized or Abdominal Edema
Description: Number of participants who had generalized or abdominal edema.
Time Frame: Baseline, Weeks 4, 20, 36, 52, and 53
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Participants
  Baseline (n=103) | 0
  Week 4 (n=101) | 0
  Week 20 (n=93) | 0
  Week 36 (n=90) | 0
  Week 52/early termination (n=100) | 1
  Week 53/early termination (n=78) | 0

4. Primary Outcome: Number of Participants With Localized Pain Related to Deep Vein Thrombosis (DVT)
Description: DVT was defined if a segment of the deep vein of the lower limb was not compressible or a previous compressive vein became non compressive or there was no flow in the underlying vessel. Symptoms of DVT included pain in the lower limb, localized tenderness, swelling, pitting edema, collateral superficial veins (non-varicose), and skin redness. The symptom was assessed as mild, moderate or severe.
Time Frame: Baseline, Weeks 4, 20, 36, 52, and 53
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Participants
  Mild at Baseline (n=103) | 2
  Moderate at Baseline (n=103) | 3
  Severe at Baseline (n=103) | 1
  Mild at Week 4 (n=101) | 5
  Moderate at Week 4 (n=101) | 1
  Severe at Week 4 (n=101) | 0
  Mild at Week 20 (n=93) | 3
  Moderate at Week 20 (n=93) | 0
  Severe at Week 20 (n=93) | 0
  Mild at Week 36 (n=90) | 3
  Moderate at Week 36 (n=90) | 0
  Severe at Week 36 (n=90) | 0
  Mild at Week 52/early termination (n=100) | 3
  Moderate at Week 52/early termination (n=100) | 0
  Severe at Week 52/early termination (n=100) | 1
  Mild at Week 53/early termination (n=78) | 2
  Moderate at Week 53/early termination (n=78) | 1
  Severe at Week 53/early termination (n=78) | 0

5. Primary Outcome: Number of Participants With Localized Tenderness Related to Deep Vein Thrombosis (DVT)
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 20, 36, 52, and 53
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Participants
  Mild at Baseline (n=103) | 0
  Moderate at Baseline (n=103) | 0
  Severe at Baseline (n=103) | 0
  Mild at Week 4 (n=101) | 0
  Moderate at Week 4 (n=101) | 0
  Severe at Week 4 (n=101) | 0
  Mild at Week 20 (n=93) | 0
  Moderate at Week 20 (n=93) | 0
  Severe at Week 20 (n=93) | 0
  Mild at Week 36 (n=90) | 0
  Moderate at Week 36 (n=90) | 0
  Severe at Week 36 (n=90) | 0
  Mild at Week 52/early termination (n=100) | 0
  Moderate at Week 52/early termination (n=100) | 0
  Severe at Week 52/early termination (n=100) | 0
  Mild at Week 53/early termination (n=78) | 0
  Moderate at Week 53/early termination (n=78) | 0
  Severe at Week 53/early termination (n=78) | 0

6. Primary Outcome: Number of Participants With Swelling Related to Deep Vein Thrombosis (DVT)
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 20, 36, 52, and 53
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Participants
  Mild at Baseline (n=103) | 4
  Moderate at Baseline (n=103) | 2
  Severe at Baseline (n=103) | 0
  Mild at Week 4 (n=101) | 3
  Moderate at Week 4 (n=101) | 2
  Severe at Week 4 (n=101) | 0
  Mild at Week 20 (n=93) | 3
  Moderate at Week 20 (n=93) | 2
  Severe at Week 20 (n=93) | 0
  Mild at Week 36 (n=90) | 4
  Moderate at Week 36 (n=90) | 1
  Severe at Week 36 (n=90) | 0
  Mild at Week 52/early termination (n=100) | 7
  Moderate at Week 52/early termination (n=100) | 0
  Severe at Week 52/early termination (n=100) | 0
  Mild at Week 53/early termination (n=78) | 5
  Moderate at Week 53/early termination (n=78) | 0
  Severe at Week 53/early termination (n=78) | 0

7. Primary Outcome: Number of Participants With Pitting Edema Related to Deep Vein Thrombosis (DVT)
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 20, 36, 52, and 53
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Participants
  Mild at Baseline (n=103) | 6
  Moderate at Baseline (n=103) | 1
  Severe at Baseline (n=103) | 0
  Mild at Week 4 (n=101) | 5
  Moderate at Week 4 (n=101) | 2
  Severe at Week 4 (n=101) | 0
  Mild at Week 20 (n=93) | 4
  Moderate at Week 20 (n=93) | 1
  Severe at Week 20 (n=93) | 0
  Mild at Week 36 (n=90) | 7
  Moderate at Week 36 (n=90) | 0
  Severe at Week 36 (n=90) | 0
  Mild at Week 52/early termination (n=100) | 8
  Moderate at Week 52/early termination (n=100) | 0
  Severe at Week 52/early termination (n=100) | 0
  Mild at Week 53/early termination (n=78) | 4
  Moderate at Week 53/early termination (n=78) | 0
  Severe at Week 53/early termination (n=78) | 0

8. Primary Outcome: Number of Participants With Collateral Superficial Veins (Non-varicose) Related to Deep Vein Thrombosis (DVT)
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 20, 36, 52, and 53
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Participants
  Mild at Baseline (n=103) | 0
  Moderate at Baseline (n=103) | 0
  Severe at Baseline (n=103) | 0
  Mild at Week 4 (n=101) | 0
  Moderate at Week 4 (n=101) | 0
  Severe at Week 4 (n=101) | 0
  Mild at Week 20 (n=93) | 0
  Moderate at Week 20 (n=93) | 0
  Severe at Week 20 (n=93) | 0
  Mild at Week 36 (n=90) | 0
  Moderate at Week 36 (n=90) | 0
  Severe at Week 36 (n=90) | 0
  Mild at Week 52/early termination (n=100) | 0
  Moderate at Week 52/early termination (n=100) | 0
  Severe at Week 52/early termination (n=100) | 0
  Mild at Week 53/early termination (n=78) | 0
  Moderate at Week 53/early termination (n=78) | 0
  Severe at Week 53/early termination (n=78) | 0

9. Primary Outcome: Number of Participants With Skin Redness Related to Deep Vein Thrombosis (DVT)
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 20, 36, 52, and 53
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Participants
  Mild at Baseline (n=103) | 0
  Moderate at Baseline (n=103) | 0
  Severe at Baseline (n=103) | 0
  Mild at Week 4 (n=101) | 0
  Moderate at Week 4 (n=101) | 0
  Severe at Week 4 (n=101) | 0
  Mild at Week 20 (n=93) | 1
  Moderate at Week 20 (n=93) | 0
  Severe at Week 20 (n=93) | 0
  Mild at Week 36 (n=90) | 0
  Moderate at Week 36 (n=90) | 0
  Severe at Week 36 (n=90) | 0
  Mild at Week 52/early termination (n=100) | 0
  Moderate at Week 52/early termination (n=100) | 0
  Severe at Week 52/early termination (n=100) | 0
  Mild at Week 53/early termination (n=78) | 0
  Moderate at Week 53/early termination (n=78) | 0
  Severe at Week 53/early termination (n=78) | 0

10. Primary Outcome: Number of Participants With Visual Field Deteriorated
Description: Number of participants who had normal visual field at baseline and showed abnormal result after the study treatment, assessed by confrontational visual field test (neurological examination).
Time Frame: 53 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Participants
  Right eye | 0
  Left eye | 0

11. Primary Outcome: Number of Participants With Deterioration in Neurological Examination Findings
Description: Worsening of the condition relative to baseline was reported as deteriorated. Assessment categories are as follows: normal or abnormal for Cranial Nerve Function, Mental State, and Coordination; normal, mild, moderate, or severe ataxia for Gait; none/absent, normal, or hyper-reflexic for Deep Tendon Reflexes; absent or present for Abnormal Reflexes; normal, mild, moderate, or severe weakness for Muscle Strength; slight, more marked, or considerable increase, or affected parts rigid in flexion or extension for Muscle Tone; absent or present for Sensory Function.
Time Frame: 53 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Participants
  Cranial Nerve Function | 0
  Mental State | 0
  Coordination: Right (R)- Finger to Nose | 0
  Coordination: Left (L)- Finger to Nose | 2
  Coordination: R- Finger Tapping | 1
  Coordination: L- Finger Tapping | 0
  Coordination: R- Rapid Alternating Hand Movement | 1
  Coordination: L- Rapid Alternating Hand Movement | 2
  Coordination: Romberg Test | 1
  Gait | 1
  Deep Tendon Reflexes: R- Brachioradialis | 1
  Deep Tendon Reflexes: L- Brachioradialis | 1
  Deep Tendon Reflexes: R-Patellar | 3
  Deep Tendon Reflexes: L-Patellar | 3
  Deep Tendon Reflexes: R- Achilles | 2
  Deep Tendon Reflexes: L- Achilles | 3
  Abnormal Reflexes | 1
  Muscle Strength: R- Upper Limb | 1
  Muscle Strength: L- Upper Limb | 2
  Muscle Strength: R- Lower Limb | 1
  Muscle Strength: L- Lower Limb | 2
  Muscle Tone: R- Upper Limb | 1
  Muscle Tone: L- Upper Limb | 1
  Muscle Tone: R- Lower Limb | 5
  Muscle Tone: L- Lower Limb | 5
  Sensory Function: Anesthesia | 0
  Sensory Function: Hypesthesia | 1
  Sensory Function: Allodynia | 1
  Sensory Function: Hyperalgesia | 2

12. Primary Outcome: Number of Participants With Suicidal Ideation According to Sheehan Suicidality Tracking Scale (Sheehan-STS)
Description: The Sheehan-STS is an 8-item prospective rating scale that tracks treatment-emergent suicidal ideation and behaviors. Participants who reported a score of ≥1 (5-point scale ranging from 0: not at all to 4: extremely) for Item 2, 3, 4 or 5 of the Sheehan-STS prognostic scale is considered to have suicidal ideation as the scores are mapped to Category 4 (suicide ideation) of the Columbia Classification Algorithm of Suicide Assessment.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 20, 28, 36, 44, and 52
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Participants
  Baseline (n=103) | 3
  Week 2 (n=102) | 2
  Week 4 (n=101) | 1
  Week 8 (n=99) | 0
  Week 12 (n=96) | 0
  Week 20 (n=93) | 2
  Week 28 (n=91) | 2
  Week 36 (n=90) | 2
  Week 44 (n=85) | 2
  Week 52 (n=101) | 0

13. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire (SF-MPQ) at Each Time Point: Total Scores
Description: The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
  Range: 0 to 45 for total score. Change = observation mean minus baseline mean. Negative change indicated improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 20, 28, 36, 44, and 52
Population: The full analysis set consists of all participants who received at least one dose of study medication in this long-term study and for whom post-treatment data were available. For study endpoint of efficacy (Week 52), missing values was imputed with the last observation carried forward (LOCF).
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Score on a scale
  Week 2 (n=103) | -4.2 [-5.4 to -3.0]
  Week 4 (n=102) | -5.2 [-6.4 to -4.0]
  Week 8 (n=99) | -5.3 [-6.6 to -4.0]
  Week 12 (n=98) | -5.7 [-7.3 to -4.2]
  Week 20 (n=95) | -6.1 [-7.6 to -4.7]
  Week 28 (n=92) | -5.1 [-6.6 to -3.6]
  Week 36 (n=91) | -5.0 [-6.5 to -3.5]
  Week 44 (n=87) | -4.4 [-6.1 to -2.8]
  Week 52 (n=85) | -5.0 [-6.6 to -3.4]
  Week 52 (LOCF, n=103) | -4.6 [-6.2 to -3.0]

14. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire (SF-MPQ) at Each Time Point: Sensory Scores
Description: The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
  Range: 0 to 33 for sensory score. Change = observation mean minus baseline mean. Negative change indicated improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 20, 28, 36, 44, and 52
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Score on a scale
  Week 2 (n=103) | -3.1 [-4.1 to -2.2]
  Week 4 (n=102) | -3.9 [-4.8 to -3.0]
  Week 8 (n=99) | -3.9 [-4.9 to -3.0]
  Week 12 (n=98) | -4.2 [-5.4 to -3.1]
  Week 20 (n=95) | -4.5 [-5.6 to -3.4]
  Week 28 (n=92) | -3.8 [-5.0 to -2.7]
  Week 36 (n=91) | -3.7 [-4.8 to -2.6]
  Week 44 (n=87) | -3.1 [-4.4 to -1.9]
  Week 52 (n=85) | -3.6 [-4.8 to -2.4]
  Week 52 (LOCF, n=103) | -3.6 [-4.8 to -2.4]

15. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire (SF-MPQ) at Each Time Point: Affective Scores
Description: The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
  Range: 0 to 12 for affective score. Change = observation mean minus baseline mean. Negative change indicated improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 20, 28, 36, 44, and 52
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Score on a scale
  Week 2 (n=103) | -1.1 [-1.5 to -0.5]
  Week 4 (n=102) | -1.3 [-1.7 to -0.8]
  Week 8 (n=99) | -1.3 [-1.8 to -0.9]
  Week 12 (n=98) | -1.5 [-2.0 to -1.0]
  Week 20 (n=95) | -1.6 [-2.1 to -1.2]
  Week 28 (n=92) | -1.3 [-1.8 to -0.9]
  Week 36 (n=91) | -1.3 [-1.8 to -0.7]
  Week 44 (n=87) | -1.3 [-1.9 to -0.7]
  Week 52 (n=85) | -1.4 [-1.9 to -0.9]
  Week 52 (LOCF, n=103) | -1.0 [-1.5 to -0.5]

16. Secondary Outcome: Change From Baseline in the Modified Brief Pain Inventory (10 Item) (mBPI-10)Total Scores at Last Evaluation Score
Description: The mBPI-10 is a self administered questionnaire that assesses pain interference with functional activities over the past week. These items are measured on an 11 point scale, ranging from "does not interfere" (0) to "completely interferes" (10). A composite score, the Pain Interference Index, will be calculated by averaging the 10 items that comprise the scale.
  Change = observation mean at Week 52 minus baseline mean.
Time Frame: Baseline, Week 52
Population: The full analysis set consists of all participants who received at least one dose of study medication in this long-term study and for whom post-treatment data were available.
  The number of participants who had mBPI at Week 52/ Early Termination was 101 participants (n=101).
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
Score on a scale | -1.4 [-1.9 to -0.9]

ADVERSE EVENTS:
Time Frame: 53 weeks
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 19/103
Other Adverse Events (participants affected / at risk) | 91/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=103)
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Tooth development disorder (Gastrointestinal disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 2
Infected skin ulcer (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Mucosal excoriation (Injury, poisoning and procedural complications) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=103)
Visual acuity reduced (Eye disorders) | 7
Constipation (Gastrointestinal disorders) | 8
Feeling abnormal (General disorders) | 7
Oedema peripheral (General disorders) | 18
Thirst (General disorders) | 7
Nasopharyngitis (Infections and infestations) | 26
Contusion (Injury, poisoning and procedural complications) | 8
Fall (Injury, poisoning and procedural complications) | 13
Weight increased (Investigations) | 31
Back pain (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 24
Hypoaesthesia (Nervous system disorders) | 6
Somnolence (Nervous system disorders) | 53
Eczema (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.